CLINICAL TRIAL: NCT06343987
Title: Feasibility of a Physical Activity Program in Patients With Metastatic Breast Cancer and Overweight: a Randomized Controlled Trial
Brief Title: The FEMA Study: Feasibility of Exercise in Patients With Metastatic Breast Cancer and Adiposity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Signe Borgquist, Chair Professor, Senior Consultant, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-165-23
Record Dates: First submitted 2024-03-06; First posted 2024-04-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Breast Cancer; Estrogen-receptor-positive Breast Cancer; Adiposity
Keywords: Metastatic Breast Cancer; Physical Activity; Adiposity; Endocrine Therapy; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Continuous inclusion. Randomized 2:1 - intervention group and observational group, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): 14 participants
  Interventions: Behavioral: Physical Activity
- Observational Arm (No Intervention): 7 participants

INTERVENTIONS:
Behavioral: Physical Activity — 12-week physical activity program with training 3 times a week. The training consists of high-intensity training such as weight-lifting and cardiovascular training, and low-intensity training such as relaxation and stretching.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to test a physical activity program in patients with metastatic breast cancer and overweight receiving endocrine-based treatment.

The aim of the study is to assess the feasibility of a 12-week physical activity program in this patient group in terms of adherence, recruitment rate, retention and acceptability. Potential effects on metabolic health, body composition, physical performance, obesity-related biomarkers and patient-related outcomes are explored. The hypothesis is that improving metabolic health and health-related quality of life through physical activity can optimize cancer care.

Participants will randomized 2:1 to either a physical activity program or care as usual.

DETAILED DESCRIPTION:
Women with overweight and obesity not only have a greater risk of developing breast cancer; they also have a worse prognosis. At diagnosis, women with overweight are more likely to have more advanced breast cancer and face an elevated risk of developing distant metastases compared to breast cancer patients with normal weight. Despite advanced disease, many patients with metastatic breast cancer can live for several years, but experience weight-gain, physical de-conditioning, and decreasing quality of life. On top of this, patients with endocrine-responsive metastatic breast cancer often receive treatment with aromatase inhibitors which can induce metabolic changes, increasing the risk of weight-gain and type 2 diabetes. The hypothesis is that improving metabolic health and quality of life through physical activity in patients with metastatic breast cancer and overweight receiving endocrine-based treatment can optimize cancer care.

Therefore, in this randomized controlled trial, the investigators will launch a 12-week physical intervention program including 21 participants to investigate the feasibility and potential effects hereof. The program will take place at Steno Diabetes Centre Aarhus, and patients are included from the Department of Oncology, Aarhus University Hospital. The physical activity program consists of training 3 times a week with a supervising physiotherapist. Throughout the study, data will be collected through blood samples, blood pressure measurements, bioelectrical impedance analysis, physical performance tests, questionnaires on quality of life, self-efficacy of cancer coping, sleep quality and a self-developed evaluation questionnaire, and one individual semi-structured interview.

This feasibility study will guide the decision of a future, full-scale study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed metastatic breast cancer
* BMI ≥ 25
* Receive first-line endocrine-based therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1

Exclusion Criteria:

* Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; these conditions will be discussed with the patient before registration in the trial.
* Physical health condition that either is unsafe for participation or prevents the patient from participating adequately in the physical activity program.
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Recruitment rate calculated by the amount of included partcipants of those eligible
Adherence to the training program | 1 year
  Adherence to the training program assessed by the mean attendance rate
Retention | 1,5 years
  Retention rate to the study assessed by the proportion of participants in each study arm that completes the study period
Adherence to other study procedures | 1,5 years
  Adherence to other study procedures assessed by the proportion of completed questionnaires and blood samples at the specified time-points
Acceptability | 1 year
  Acceptability of the study intervention assessed by the proportion of participants in the intervention arm that anwers "yes" to the question: "Would you recommend others to participate in the physical activity program?"

OTHER OUTCOMES:
Health-related quality of life as assessed by EORTC-QLQ-30 | Until the end of study
  Change in health-related quality of life measured with European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status/QoL scale, and six single items, with 30 items in total. All scales and single-item measures range in score from 0 to 100. A high score on the functional scale represents a high level of functioning, a high score for the global health status represents a high HRQoL, but a high score on a symptom scale represents a high level of symptomatology
Metabolic score | Until the end of study
  Change in metabolic score calculated as the sum of Z-transformed levels of mid-blood pressure [(systolic blood pressure + diastolic blood pressure)/2], glucose, and triglycerides. A higher score indicates a worse metabolic health
Self-efficacy of cancer coping as assessed by CBI-12 | Until end of study
  Change in self-efficacy in coping with cancer measured with Cancer Behavior Inventory-12 (CBI-12). The questionnaire is scored as a one-dimensional scale, summing the ratings for the items. A higher score indicates higher levels of self-efficacy, with a maximum score of 108.
Sleep quality as assessed by PSQI | Until end of study
  Change in sleep quality measured with Pittsburgh Sleep Quality Index (PSQI). The questionnaire consists of 19 items grouped into seven component scores. The directionality and interpretation of scores vary across items. A total score ranging from 0 to 21 can be calculated, with a higher score indicating poorer sleep quality. A score < 5 indicates good sleep quality.
Insomnia as assessed by ISI | Until end of study
  Change in insomnia assessed by Insomnia Severity Index (ISI). It contains 7 items and is scored on a one-dimensional scale with a maximum score of 28. The total score is grouped into four categories: no insomnia (0-7), subclinical insomnia (8-14), clinical insomnia (15-21) and severe clinical insomnia (22-28).
Change in C-reactive protein | 1 year
  Change in circulation levels of C-reactive protein measured in mg/L
Change in leukocytes | 1 year
  Change in circulation levels of total leukocytes measured in 10^9/L
Change in HbA1c | 1 year
  Change in HbA1c measured in mmol/mol
Change in LDL cholesterol | 1 year
  Change in LDL cholesterol measured in mmol/L
Change in HDL cholesterol | 1 year
  Change in HDL cholesterol measured in mmol/L
Change in BMI | 1 year
  Change in BMI kg/m^2
Fat mass | 1 year
  Change in fat mass in kilogram
Muscle mass | 1 year
  Change in muscle mass in kilogram
Visceral fat | 1 year
  Change in visceral fat in kilogram
VO2 max | 1 year
  Change in VO2 max measured by Watt-Max test
Handgrip strength | 1 year
  Change in handgrip strength in kilogram measured by dynamometer after 12 weeks
Sit-rising | 1 year
  Change in number of performed sit-rising in 30 seconds measured through a sitting-rising test

CONTACTS AND LOCATIONS:
Overall Officials: Signe SB Borgquist, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Oncology, Aarhus University Hospital, Aarhus N, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wissing M, Skovlund P, Drysdale S, Amidi A, Zachariae R, Laurberg T, Borgquist S. Feasibility of an exercise program in endocrine-treated metastatic breast cancer patients with overweight: protocol for the FEMA study. Pilot Feasibility Stud. 2025 Apr 2;11(1):36. doi: 10.1186/s40814-025-01621-9. PMID 40176194